CLINICAL TRIAL: NCT00760253
Title: Compare the Side Effects and Differences Awake Level of Propofol by Using Three TCI Formula of Anesthesia in TVOR Patients
Brief Title: Compare the Side Effects and Difference Awake Level of Three TCI Propofol Formula in TVOR Patients
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Jeng Chuen-shin/ visiting staff of Anesthesiology, NTUH, NTUH
Other Study IDs: 200807070R
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2008-12

CONDITIONS: Bispectral Index; Transcutaneous Carbon Dioxide; PONV; Blood Pressure; Heart Rate
Keywords: target control infusion; alfentanyl; propofol; BIS
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: pure propofol by TCI pump with titration.
- 2: 10ug/kg alfentanyl bolus and propofol TCI pump infusion with titration
- 3: 20ug/kg alfentanyl bolus and propofol TCI pump infusion with titration

SUMMARY:
This study is to find the fewer side effects formula of anesthesia for TVOR patients, to compare the BIS level during emergence and to find the correlation between BIS and transcutaneous carbon dioxide concentration.

DETAILED DESCRIPTION:
Transvaginal oocyte retrieval (TVOR) is a procedure often used in infertility women . During the procedure, sedation, analgesia or anesthesia are often required. Propofol and alfentanyl are used for these patients for years, but these drugs are used in intravenous form and can be found in follicular fluid. Although further investigation needs to be undertaken to investigate any potential influence on fertilization and implantation rates, we anesthesiologist want to lower the use of drugs in these women. Target-controlled infusion (TCI) pumps can estimate and calculate the target and plasma concentration of propofol. By using these pumps , we can estimate the stable concentration of drugs. Besides, Bispectral index (BIS) monitor can help us to evaluate awareness or unarousable amnesia when we turn lower the drug use and keep patients amnesia during the procedure. Transcutaneous carbon dioxide monitor (tcCO2) can mimic the level of CO2 in patients by using noninvasive method. During anesthesia, CO2 will retain and may induce CO2 nacrosis, so we use these noninvasive method to help us to detect CO2 level preventing CO2 nacrosis and to see if there are any relationship with BIS.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II women age between 25 and 45 y/o participating to receive TVOR

Exclusion Criteria:

* Allergy history to alfentanyl, propofol or lidocaine

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: ASA physical status I or II women age between 25 and 45 y/o participating to receive TVOR procedure.
Sampling Method: Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Vital signs changes and side effects of drugs among groups | pre-anesthesia, post-anesthesia, and one hour post-anesthesia

SECONDARY OUTCOMES:
Correlation between transcutaneous carbon dioxide and BIS (bispectral index) | From drug infusion stopped to patients awake (per minute)

CONTACTS AND LOCATIONS:
Overall Officials: Chuen-shin Jeng, MD, MS, Study Director — Visiting staff
Locations (1):
- Department of Anesthesiology, National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Sherry E. Admixture of propofol and alfentanil. Use for intravenous sedation and analgesia during transvaginal oocyte retrieval. Anaesthesia. 1992 Jun;47(6):477-9. doi: 10.1111/j.1365-2044.1992.tb02268.x. PMID 1616081
- [Background] Eger EI, White PF, Bogetz MS. Clinical and economic factors important to anaesthetic choice for day-case surgery. Pharmacoeconomics. 2000 Mar;17(3):245-62. doi: 10.2165/00019053-200017030-00003. PMID 10947300
- [Background] Handa-Tsutsui F, Kodaka M. Effect of nitrous oxide on propofol requirement during target-controlled infusion for oocyte retrieval. Int J Obstet Anesth. 2007 Jan;16(1):13-6. doi: 10.1016/j.ijoa.2006.08.001. Epub 2006 Nov 27. PMID 17125991
- [Background] Soussis I, Boyd O, Paraschos T, Duffy S, Bower S, Troughton P, Lowe J, Grounds R. Follicular fluid levels of midazolam, fentanyl, and alfentanil during transvaginal oocyte retrieval. Fertil Steril. 1995 Nov;64(5):1003-7. PMID 7589618
- [Background] Chhajed PN, Rajasekaran R, Kaegi B, Chhajed TP, Pflimlin E, Leuppi J, Tamm M. Measurement of combined oximetry and cutaneous capnography during flexible bronchoscopy. Eur Respir J. 2006 Aug;28(2):386-90. doi: 10.1183/09031936.06.00088005. Epub 2006 Apr 26. PMID 16641122
- [Background] Turnbull D, Furlonger A, Andrzejowski J. The influence of changes in end-tidal carbon dioxide upon the Bispectral Index. Anaesthesia. 2008 May;63(5):458-62. doi: 10.1111/j.1365-2044.2007.05399.x. PMID 18412642
- [Background] Rigouzzo A, Girault L, Louvet N, Servin F, De-Smet T, Piat V, Seeman R, Murat I, Constant I. The relationship between bispectral index and propofol during target-controlled infusion anesthesia: a comparative study between children and young adults. Anesth Analg. 2008 Apr;106(4):1109-16, table of contents. doi: 10.1213/ane.0b013e318164f388. PMID 18349180
- [Background] Wang LP, McLoughlin P, Paech MJ, Kurowski I, Brandon EL. Low and moderate remifentanil infusion rates do not alter target-controlled infusion propofol concentrations necessary to maintain anesthesia as assessed by bispectral index monitoring. Anesth Analg. 2007 Feb;104(2):325-31. doi: 10.1213/01.ane.0000252966.03103.89. PMID 17242088
- [Background] Jeleazcov C, Ihmsen H, Schmidt J, Ammon C, Schwilden H, Schuttler J, Fechner J. Pharmacodynamic modelling of the bispectral index response to propofol-based anaesthesia during general surgery in children. Br J Anaesth. 2008 Apr;100(4):509-16. doi: 10.1093/bja/aem408. Epub 2008 Feb 12. PMID 18270231